CLINICAL TRIAL: NCT06973265
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Pain, Lymphedema, Upper Extremity Functions, and Quality of Life in Patients Undergoing Breast Surgery After Neoadjuvant Chemotherapy
Brief Title: Effects of Transcutaneous Electrical Nerve Stimulation on Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seda Akutay (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Seda Akutay, Director, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUniversity
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Surgery; Transcutaneous Electric Nerve Stimulation
Keywords: pain; lymphedema; Mastectomy; Mobility Limitation; Quality of Life
MeSH Terms: conditions — Pain; Lymphedema; Mobility Limitation | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: TENS group and control group
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS group (Experimental): Patients in this group will receive TENS treatment for 1 month after surgery.
  Interventions: Device: TENS
- Control group (No Intervention): Patients in this group do not receive TENS application after surgery.

INTERVENTIONS:
Device: TENS — After the surgery, 2 TENS electrodes will be placed on the inner part of the upper arm of the patient's arm on the side where surgery was performed, and the frequency will be 100 Hz, the pulse duration will be 100 µs and the amplitude will be adjusted so as not to cause muscle contraction, and a 20-minute TENS application will be performed.
  Arms: TENS group

SUMMARY:
The aim of this randomized controlled trial was to evaluate the effects of transcutaneous electrical nerve stimulation (TENS) on postoperative pain, lymphedema development, shoulder range of motion, and quality of life in women undergoing breast cancer surgery after neoadjuvant chemotherapy. The main questions it aims to answer are:

Does TENS reduce postoperative pain? Does TENS prevent postoperative lymphedema? Does TENS increase postoperative shoulder range of motion? Does TENS improve postoperative quality of life? The researchers will compare the effects of TENS after breast surgery with a control group.

Participants will be assessed for pain, lymphedema development, and shoulder range of motion before surgery, on the first day after surgery, at the first month after surgery, and at the third month after surgery. Quality of life will be assessed before surgery, at the first month after surgery, and at the third month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Those whose primary cancer tissue is breast
* ASA classification is between I and III
* Having unilateral breast surgery

Exclusion Criteria:

* Those with cardiac problems and those using a pacemaker
* Pregnant
* Cognitively impaired
* Disruption of skin integrity in the TENS application area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Until the end of 3 month
  The Visual Analog Scale (VAS) scale will be used to assess pain intensity. It is a 10 cm line with connecting expressions on the left (no pain) and on the right (extreme pain). The patient is asked to mark the current pain level on the line. It means that the pain intensity increases as you move from left to right.
Lymphedema severity | Until the end of 3 month
  A tape measure will be used to assess the severity of lymphedema. Measurements will be made bilaterally at 6 different points (Hand circumference, wrist, 15 cm below the elbow, 7,5 cm below the elbow, 7,5 cm above the elbow, 15 cm above the elbow )on the arm.
Shoulder and arm mobility | Until the end of 3 month
  Shoulder range of motion (flexion, extension, abduction, internal rotation and external rotation angles of the arm) was measured with a goniometer.

SECONDARY OUTCOMES:
Upper extremity functions | Preoperative period, postoperative 1 month and postoperative 3 month
  The Quick Disability of the Arm, Shoulder and Hand (QuickDASH) Questionnaire and hand dynamometer will be used. In QuickDASH, a higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability.
Cancer Related Quality of Life | Preoperative period, postoperative 1 month and postoperative 3 month
  European Organization for Cancer Research and Treatment Quality of Life Questionnaire-30- EORTC QLQ-C30 will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akutay S, Yuceler Kacmaz H, Ceyhan O. The healing power of transcutaneous electrical nerve stimulation: a systematic review on its effects after breast surgery. Support Care Cancer. 2025 Jan 13;33(2):90. doi: 10.1007/s00520-024-09129-3. PMID 39804405